CLINICAL TRIAL: NCT03315221
Title: Renoir: A Randomised, Double-blind, Controlled Trial to Evaluate the Effects of a New Human Milk Fortifier on Growth and Tolerance in Preterm Infants.
Acronym: Renoir
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EBB16GL06402
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Subjects in Need of a Human Milk Fortifier (HMF); Growth; Tolerance; Safety
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): Human Milk Fortifier (HMF) with added lipids.
  Interventions: Other: Test product
- Control product (Active Comparator): Commercially available HMF (without lipids).
  Interventions: Other: Control product

INTERVENTIONS:
Other: Test product — HMF with added lipids - Intervention group
  Arms: Test product
Other: Control product — Commercially available HMF (without lipids) - control group
  Arms: Control product

SUMMARY:
Preterm birth (birth before start of the 37th week of gestation) is a major determinant of neonatal morbidity and mortality and has long-term adverse consequences for health and neurodevelopment.

Preterm infants have much higher nutrient requirements than term infants. The preferred nutrition for all infants including preterm infants is human milk from the infant's own mother, or alternatively donor human milk, provided it is fortified with several nutrients as human milk alone does not sufficiently meet the nutritional needs of preterm infants.

Human milk fortifiers (HMFs) are multicomponent enrichments that can be added to human milk (own mother´s milk or donor milk) to meet the increased nutritional needs of preterm infants. The current Nutricia HMF (control product) has been available in its current composition since 2010. It is a multicomponent HMF providing protein, energy, minerals, and vitamins in accordance with the ESPGHAN recommendations.

Recent investigation suggests positive effects on growth and development of preterm infants when lipids are added to their nutrition. Therefore, Nutricia has added lipids to their HMF (test product) for a nutritionally more complete fortification of human milk aiming for optimal growth and optimal cognitive and brain development.

The Renoir study will investigate the difference between both HMFs with regards to the growth velocity as well as the safety and tolerance of the new HMF.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants fed own mother's milk (or donor human milk) in need of a HMF (as decided by the investigator)
2. Gestational age <32 weeks and birth weight <1500 g
3. Receiving enteral feeding
4. Expected to need a HMF for minimally 21 days
5. Written informed consent from custodial parent(s)

Exclusion Criteria:

1. Any relevant proven or suspected chromosomal anomaly, metabolic disorder, genetic syndrome or congenital central nervous system malformation;
2. Presence or history of any gastrointestinal malformation, including Necrotising enterocolitis (NEC) (defined as Bell's stage two or higher);
3. No realistic prospect of survival at the discretion of the attending physician;
4. Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study;
5. Expected or foreseen inability of the subject and/or their families to adhere to protocol instructions.

Ages: 1 Week to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Weight growth velocity | 21 days
  Weight growth velocity (in g/kg/day) from baseline to study day 21

SECONDARY OUTCOMES:
Length | up to 16 weeks, depending on gestational age at birth
  Length gain (cm/week)
Head circumference | up to 16 weeks, depending on gestational age at birth
  Head circumference gain (cm/week)
Weight for Length | up to 16 weeks, depending on gestational age at birth
  Weight for Length
Z-scores | up to 16 weeks, depending on gestational age at birth
  Z-scores (no unit) of anthropometric measures (weight for age, length for age, head circumference for age)
Stool consistency | up to 16 weeks, depending on gestational age at birth
  Stool consistency (4-point scale Amsterdam stool scale: watery, soft, formed, hard)
Stool frequency | up to 16 weeks, depending on gestational age at birth
  Stool frequency (number of stools per day)
Enteral intake | up to 16 weeks, depending on gestational age at birth
  Total enteral intake (mL/kg/day)
vomiting | up to 16 weeks, depending on gestational age at birth
  Incidence of vomiting (number/day)
Regurgitation | up to 16 weeks, depending on gestational age at birth
  Incidence of regurgitation (number/day)
Enteral feed | up to 16 weeks, depending on gestational age at birth.
  Number of days that an infant is not fed enterally

OTHER OUTCOMES:
Exploratory - Age | 2-16 weeks, depending on gestational age at birth
  Age at discharge from the neonatal intensive care unit (NICU, level III)
Exploratory - Age | 4-16 weeks depending on gestational age at birth
  Age at discharge home
Exploratory - Mortality | up to 16 weeks depending on gestational age at birth
  Mortality (yes/no) during stay in NICU/hospital
Exploratory - Enteral feeding volume | around 1-4 weeks, depending on gestational age at birth
  Time in days to achieve an enteral feeding volume of at least 150 mL/kg/day +/- 10 mL for 3 consecutive days
Exploratory - Gastric residuals | up to 16 weeks, depending on gestational age at birth
  Frequency of clinically significant gastric residuals, defined as gastric residuals leading to a change in feeding according to the investigator's assessment (if assessed per local standard practice)
Exploratory - Diarrhoea | up to 16 weeks, depending on gestational age at birth)
  Occurrence of diarrhoea
Exploratory - Constipation | up to 16 weeks, depending on gestational age at birth)
  Occurrence of constipation
Exploratory - Weight | at 6, 12 and 24 months corrected age (CA)
  Weight (g)
Exploratory - Length | at 6, 12 and 24 months corrected age (CA)
  Length (cm)
Exploratory - Head circumference | at 6, 12 and 24 months corrected age (CA)
  Head circumference (cm)
Exploratory - Neurodevelopmental outcome | at 24 months CA
  Neurodevelopmental outcome assessed by Bayley Scales of Infant and Toddler Development, Third Edition, on three subscales (cognitive, fine and gross motor)
Safety - Incidence (S)AE's | up to 24 months CA
  Incidence of (Serious) Adverse Events that are assessed by the Investigator to be possibly, probably or definitely related to the study product
Safety - Frequency (S)AE's | up to 24 months CA
  Frequency of (Serious) Adverse Events that are assessed by the Investigator to be possibly, probably or definitely related to the study product
Safety - Severity (S)AE's | up to 24 months CA
  Severity of (Serious) Adverse Events (mild/moderate/severe) that are assessed by the Investigator to be possibly, probably or definitely related to the study product
Safety - Relatedness (S)AE's | up to 24 months CA
  Relatedness of Serious Adverse Events
Safety - Incidence Blood in stool | up to 16 weeks, depending on gestational age at birth)
  Incidence blood in stool
Safety - Frequency Blood in stool | up to 16 weeks, depending on gestational age at birth)
  Frequency of blood in stool
Safety - Severity Blood in stool | up to 16 weeks, depending on gestational age at birth)
  Severity of blood in stool (mild, moderate, severe)
Safety - NEC | up to 16 weeks, depending on gestational age at birth)
  NEC (defined as Bell's stage two or higher) (as part of the assessment of neonatal morbidity)
Safety - Bronchopulmonary dysplasia | up to 16 weeks, depending on gestational age at birth)
  Bronchopulmonary dysplasia (as part of the assessment of neonatal morbidity), categorized into mild/moderate/severe based on Sahni et al
Safety - Serious neonatal infections | up to 16 weeks, depending on gestational age at birth
  Serious neonatal infections (as part of the assessment of neonatal morbidity), i.e. confirmed sepsis, pneumonia, or meningitis
Safety - Retinopathy of Prematurity | up to 16 weeks, depending on gestational age at birth
  Retinopathy of Prematurity, based on International Committee for the Classification of Retinopathy of Prematurity (as part of the assessment of neonatal morbidity)
Safety - Metabolic acidosis | up to 16 weeks, depending on gestational age at birth
  Metabolic acidosis (as part of the assessment of neonatal morbidity) leading to correction and/or change in clinical management of the subject (according to the investigator's assessment)

CONTACTS AND LOCATIONS:
Locations (15):
- France (2):
  - Hôpital de la Croix Rousse, Lyon
  - CHRU Nancy - Maternité regionale Universitaire A. Pinard, Nancy
- Germany (2):
  - Universitätskinderklinik der Otto-v.-Guericke Universität, Magdeburg
  - Klinikum Nürnberg Süd, Nuremberg
- Netherlands (9):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - Flevoziekenhuis, Almere Stad
  - Amsterdam UMC (VUMC), Amsterdam
  - OLVG Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Spaarne Ziekenhuis, Hoofddorp
  - Maastricht UMC, Maastricht
  - VieCuri Medisch Centrum, Venlo
  - Isala Ziekenhuis, Zwolle
- United Kingdom (2):
  - Saint-Peter's Hospital NHS Foundation Trust, Chertsey
  - Norfolk and Norwich NHS Foundation Trust, Norwich

REFERENCES:
- [Derived] Picaud JC, Reynolds PR, Clarke P, van den Hooven E, van Weissenbruch MM, van Lingen RA, Goedhart A, Botma A, Boettger R, van Westering-Kroon E, Fusch C, Hascoet JM; RENOIR Study Group. A novel human milk fortifier supports adequate growth in very low birth weight infants: a non-inferiority randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2025 Aug 19;110(5):512-519. doi: 10.1136/archdischild-2024-327282. PMID 40037774